CLINICAL TRIAL: NCT05466565
Title: Exploratory Study on Optimized Antiviral Strategy After Radical Resection of Hepatitis B-related Hepatocellular Carcinoma
Brief Title: Antiviral Therapy for Patients With Liver Cancer After Surgery
Status: Recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: XiangyaHGRS
Record Dates: First submitted 2022-07-18; First posted 2022-07-20 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Radical Surgery for Liver Cancer; antiviral therapy
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Nucleoside analog alone group: planning or ongoing treatment with entecavir (ETV), tenofovir disoproxil fumarate (TDF), tenofovir alafenamide (TAF), and no addition or switch Patients on the pegylated interferon alfa-2b program
- In the continuous treatment group of peginterferon: the subjects started oral antiviral drugs from the 2nd day after operation, and simultaneously took peginterferon alfa-2b in combination from the 4th to 8th week after operation, and stopped after 96 weeks. Continue oral antiviral drugs with peginterferon
- In the pegylated interferon pulse medication group: the subjects started oral antiviral drugs from the second day after the operation, and at any time point from the 4th to the 8th week after the operation, the subjects were combined with peginterferon alfa-2b. After every 8 weeks of combined use, stop for 4 weeks (continuous oral NA is maintained during the period), and perform periodically until pegylated interferon is stopped after 96 weeks, and oral antiviral drugs are continued

SUMMARY:
This is a single-center, prospective, observational, real world study designed to evaluate the effects of peginterferon α-2b(pegabin) combined with nucleoside (acid) analogs (entecavir,ETV tenofovir,TDF tenofovir alafenamide,TAF) on patients after radical surgery for hepatitis B associated hepatocellular carcinoma by collecting data from patients at our hospital

DETAILED DESCRIPTION:
In this study, patients eligible for conventional oral antiviral therapy (ETV, TDF and TAF) after radical surgery for HBV-HCC will be screened, and the subjects who fully meet the inclusion and exclusion criteria will be included in the study after signing the informed consent letter according to the different treatment regiments received by the patients. Baseline information will be collected and relevant test and examination data will be collected at fixed time points after the initiation of treatment. Enrolled patients will be divided into three groups according to treatment regiments: GROUP A, group B and group C. Each group is expected to include 120 subjects, and A total of 360 subjects will be collected Group A: patients in the nucleoside analogues alone group who planned or were receiving entecavir (ETV) tenofovir fumarate (TDF) propofol tenofovir fumarate (TAF) and did not add or switch to peg interferin A-2B program Group B: peG-interferon continuous administration group, subjects were given oral antiviral drugs from day 2 after surgery, and peg-interferon α-2b was combined with peg-interferon α -2B from week 4 to 8 after surgery, until peg-interferon was stopped and antiviral drugs were continued after 96 weeks Group C: polyethylene glycol interferon pulse treatment group, the subjects since 2 days after oral antiviral drugs, at the same time of 4 to 8 week after any point in time with polyethylene glycol interferon alpha 2 b, 8 weeks after stopping each combination (keep continuous oral NA) during 4 weeks, periodic, until weeks after stop using polyethylene glycol (peg) 96 interferon, continue to oral antiviral drugs Follow the instructions for oral antiviral drug administration Patients returned to the study center at weeks 4, 8, 12, 24, 36, 48, 60, 72, 84, 96, and every 12 weeks thereafter, with a 7-day treatment window and a 15-day follow-up window, until 5 years or study termination Regardless of the reason for discontinuing the study drug therapy, the investigator should try to persuade the patient to continue to complete the 5-year survival follow-up and collect the following information: patient survival status and subsequent treatment options (including targeted therapy, chemotherapy, radiotherapy, surgery and immunotherapy) The primary outcome measures were recurrence free survival (RFS), and the secondary outcome measures were the decrease of HBsAg relative to baseline and the dynamic change of cccDNA clearance rate (OS), which could be used to comprehensively compare the efficacy of combined treatment with peginterferon α-2b after radical surgery

ELIGIBILITY:
Inclusion Criteria:

* 1. Age: 18-65 years old, gender is not limited; 2. Patients with hepatocellular carcinoma after radical surgical resection or radiofrequency ablation; 3. HBsAg positive; 4. Intraoperative pathology showed no residual incision margin, and imaging confirmed as complete remission (CR) within 4 weeks after operation; 5. The investigator evaluates that they can receive peginterferon and nucleoside (acid) analog therapy; 6. Sign the informed consent form and be able to comply with the requirements of the program; if the patient cannot sign the informed consent form, his/her legal guardian or agent must sign it.

Exclusion Criteria:

* 1. Are receiving hepatotoxic drugs, immunosuppressants or targeted drug therapy, or receiving adjuvant chemotherapy after surgery; 2. Past or concurrent with other malignant tumors, except for cured skin basal cell or squamous cell carcinoma and cervical carcinoma in situ; 3. Those who are allergic to interferon alpha and its drug components, and those who are judged by the investigator to be unsuitable for the use of interferon alpha; 4. Combined with HAV, HCV, HDV, HEV, HIV infection, alcoholic liver disease, genetic metabolic liver disease, drug-induced liver disease, non-alcoholic fatty liver disease and other chronic liver diseases; combined with autoimmune diseases, including autoimmune liver disease, Psoriasis, etc.; 5. Neutrophil count < 1.5 x 109 cells/L or platelet count < 80 x 109 cells/L; 6. Creatinine is higher than 1.5 times the upper limit of normal; 7. Patients with serious diseases of the heart, lung, kidney, brain, blood and other important organs; 8. Patients with severe neurological and psychiatric diseases (such as epilepsy, depression, mania, seizures, schizophrenia, etc.); 9. Unstable control of diabetes, hypertension, thyroid disease, etc.; history of severe retinopathy or patients with retinopathy shown by other evidence; 10. Child-Pugh is graded C; 11. Drug abuse or alcoholism; 12. Infection, hemorrhage or other postoperative complications deemed unsuitable to participate in the study during the baseline examination; the baseline examination indicates the recurrence and metastasis of liver cancer; 13. Pregnant or breastfeeding women or patients who have a pregnancy plan and are unwilling to contracept during the study period; 14. The investigator believes that the subject's current condition is not suitable for participating in this study; 15. Patients who participate in other clinical research trials at the same time.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Postoperative hepatocellular carcinoma patients with chronic hepatitis B
Sampling Method: Non-Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
recurrence-free survival time | 240 weeks
  no new liver cancer

SECONDARY OUTCOMES:
Overall survival (OS) | 240 weeks
  Overall survival time of patients after radical resection of liver cancer
HBsAg reduction relative to baseline | 240 weeks
  Changes of HBsAg after antiviral therapy
Dynamic changes of cccDNA | 240 weeks
  Changes of cccDNA content in stem cells

CONTACTS AND LOCATIONS:
Overall Officials: Ledu Zhou, PhD student, Study Chair — Xiangya Hospital of Central South University
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: End of study
Access Criteria: Editors and reviewers of contributing magazines